CLINICAL TRIAL: NCT00200629
Title: A Pilot Study Examining the Value of Combined Exercise and Adenosine Stress Myocardial Perfusion Imaging as Compared With Adenosine Testing Alone for the Evaluation of Women at Intermediate or High Likelihood for Coronary Artery Disease
Brief Title: Both Exercise and Adenosine Stress Testing
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: Midwest Heart Foundation (Other)
Collaborators: GE Healthcare (Industry); Astellas Pharma US, Inc. (Industry)
Responsible Party: Kathleen Franke, Midwest Heart Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SPEC-BB
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2011-08-09 (Estimated); Status verified 2011-08

CONDITIONS: Coronary Artery Disease
Keywords: Women; Diagnostic Testing; Radionuclide Imaging; Stress Testing; Adenosine
MeSH Terms: conditions — Coronary Artery Disease

INTERVENTIONS:
Procedure: Adenosine SPECT myocardial perfusion imaging
Procedure: Combined adenosine / exercise SPECT myocardial perfusion imaging

SUMMARY:
The purpose of this study is to compare the 2-year cardiac outcomes for women with limited exercise capability based on the resuls of either pharmacological stress myocardial perfusion imaging or a combined protocol that incorporates both exercise and pharmacological stress. The goal of the study is to compare these two methods for patient tolerability, safety and prognostic value

DETAILED DESCRIPTION:
Coronary artery disease remains the leading cause of morbidity and mortality in women accounting for more than 250,000 deaths per year. Despite the high prevalence in ischemic heart disease in women, most clinical trials have focused on male cohorts. The optimal non-invasive test for evaluation of ischemic heart disease in women is unknown. A number of different modalities have been employed including exercise ECG stress testing, 2-dimensional stress echocardiography, SPECT myocardial perfusion imaging, and electron beam computerized tomography.

The cohort of women for whom to perform testing upon is also ill-defined. Myocardial perfusion imaging, in conjunction with pharmacologic stress testing, has also been shown to be effective in the diagnosis of women with known or suspected coronary artery disease as well as in for risk stratification. Recently, pharmacologic stress has been combined with low-level exercise, enhancing test tolerability and SPECT perfusion image quality. Furthermore, the use of a combined adenosine and exercise protocol may detect greater amounts of ischemia with perfusion imaging that with an exercise test alone. Therefore, in women who may be unable to perform maximal exercise, this combined pharmacologic and exercise imaging protocol may possess a significant advantage over adenosine stress testing alone.

The aim of this study is to compare safety and symptoms associated with these two methods of stress testing. The current study also seeks to establish the optimal method for detection of coronary artery disease in women who have a limited capacity for exercise (DASI score ≤5 METS), also well as examine the prognostic value of each method of testing by comparing the two-year event rates for women who undergo adenosine SPECT imaging or SPECT imaging using adenosine with adjunctive exercise.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age greater to or equal to 60 years old
* Must present with chest pain, fatigue, or other anginal equivalent symptoms
* Must be referred for stress testing based on clinical indications
* Must be able to provide written informed consent

Exclusion Criteria:

* Women with known coronary artery disease (>50% lesion OR prior MI OR prior revascularization)
* Inability to perform any exercise on a treadmill
* Nuclear medicine study within the preceding 30 days
* Contraindication to adenosine, including moderate to severe COPD or asthma, second or third degree AV block, or known hypersensitivity to adenosine or aminophylline
* Left bundle branch block or electronic ventricular pacemaker
* Significant valvular heart disease
* Hemodynamic instability (blood pressure >210/110 ml/Hg or <90/60 mm/Hg)
* 2° or 3° atrioventricular block
* Symptomatic heart failure
* Ingestion of theophylline or dipyridamole within the preceding 48 hours
* Unavailability for follow-up

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2005-06

PRIMARY OUTCOMES:
Unstable angina requiring hospitalization
non-fatal myocardial infarction
death (cardiac and noncardiac)
stroke
performance of PCI or CABG if more than 1 month after initial evaluation
hospitalization for heart failure after initial treatment is administered.

SECONDARY OUTCOMES:
Quality of Life measures (assessed by Duke Activity Status Index and Seattle Angina Questionnaire) at 6, 12, 18, and 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hendel, MD, Principal Investigator — Midwest Heart Foundation
Locations (19):
- United States (19):
  - Southwest Heart, Tucson, Arizona
  - Sutter Roseville Medical Center, Roseville, California
  - Sacramento Heart & Vascular Research Center, Sacramento, California
  - Delaware SPECT Imaging, Newark, Delaware
  - Diagnostic Cardiology, PA, Jacksonville, Florida
  - Jacksonville Heart Center, PA, Jacksonville Beach, Florida
  - Cardiac Disease Specialists, Atlanta, Georgia
  - Idaho Cardiology Associates, Boise, Idaho
  - Idaho Cardiology Associates, Meridian, Idaho
  - North Shore Cardiology, Bannockburn, Illinois
  - Iowa Heart Center, Des Moines, Iowa
  - Androscoggin Cardiology Associates, Auburn, Maine
  - Cardiovascular Consultants of Maine, PA, Scarborough, Maine
  - Albany Associates in Cardiology, Albany, New York
  - Mid-Valley Cardiology, Kingston, New York
  - North Shore University Hospital, Manhasset, New York
  - Cardiology Consultants of Philadelphia, Philadelphia, Pennsylvania
  - Medical University of SC, Charleston, South Carolina
  - Deaconess Medical Center, Spokane, Washington

REFERENCES:
- [Background] American Heart Association. 2002 Heart and Stroke Statistical Update. Dallas, Texas: American Heart Association; 2002.
- [Background] Mieres JH, Shaw LJ, Hendel RC, Miller DD, Bonow RO, Berman DS, Heller GV, Mieres JH, Bairey-Merz CN, Berman DS, Bonow RO, Cacciabaudo JM, Heller GV, Hendel RC, Kiess MC, Miller DD, Polk DM, Shaw LJ, Smanio PE, Walsh MN; Writing Group on Perfusion Imaging in Women. American Society of Nuclear Cardiology consensus statement: Task Force on Women and Coronary Artery Disease--the role of myocardial perfusion imaging in the clinical evaluation of coronary artery disease in women [correction]. J Nucl Cardiol. 2003 Jan-Feb;10(1):95-101. doi: 10.1067/mnc.2003.130362. No abstract available. PMID 12569338
- [Background] Shaw LJ, Miller DD, Romeis JC, Kargl D, Younis LT, Chaitman BR. Gender differences in the noninvasive evaluation and management of patients with suspected coronary artery disease. Ann Intern Med. 1994 Apr 1;120(7):559-66. doi: 10.7326/0003-4819-120-7-199404010-00005. PMID 8116993
- [Background] Mosca L, Grundy SM, Judelson D, King K, Limacher M, Oparil S, Pasternak R, Pearson TA, Redberg RF, Smith SC Jr, Winston M, Zinberg S. Guide to Preventive Cardiology for Women.AHA/ACC Scientific Statement Consensus panel statement. Circulation. 1999 May 11;99(18):2480-4. doi: 10.1161/01.cir.99.18.2480. No abstract available. PMID 10318674
- [Background] Holdright DR, Fox KM. Characterization and identification of women with angina pectoris. Eur Heart J. 1996 Apr;17(4):510-7. doi: 10.1093/oxfordjournals.eurheartj.a014902. No abstract available. PMID 8733082
- [Background] Gibbons RJ, Balady GJ, Beasley JW, Bricker JT, Duvernoy WF, Froelicher VF, Mark DB, Marwick TH, McCallister BD, Thompson PD, Winters WL Jr, Yanowitz FG, Ritchie JL, Cheitlin MD, Eagle KA, Gardner TJ, Garson A Jr, Lewis RP, O'Rourke RA, Ryan TJ. ACC/AHA guidelines for exercise testing: executive summary. A report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Committee on Exercise Testing). Circulation. 1997 Jul 1;96(1):345-54. doi: 10.1161/01.cir.96.1.345. No abstract available. PMID 9236456
- [Background] Hlatky MA, Pryor DB, Harrell FE Jr, Califf RM, Mark DB, Rosati RA. Factors affecting sensitivity and specificity of exercise electrocardiography. Multivariable analysis. Am J Med. 1984 Jul;77(1):64-71. doi: 10.1016/0002-9343(84)90437-6. PMID 6741986
- [Background] Kwok Y, Kim C, Grady D, Segal M, Redberg R. Meta-analysis of exercise testing to detect coronary artery disease in women. Am J Cardiol. 1999 Mar 1;83(5):660-6. doi: 10.1016/s0002-9149(98)00963-1. PMID 10080415
- [Background] Iskandrian AE, Heo J, Nallamothu N. Detection of coronary artery disease in women with use of stress single-photon emission computed tomography myocardial perfusion imaging. J Nucl Cardiol. 1997 Jul-Aug;4(4):329-35. doi: 10.1016/s1071-3581(97)90111-2. No abstract available. PMID 9278880
- [Background] Santana-Boado C, Candell-Riera J, Castell-Conesa J, Aguade-Bruix S, Garcia-Burillo A, Canela T, Gonzalez JM, Cortadellas J, Ortega D, Soler-Soler J. Diagnostic accuracy of technetium-99m-MIBI myocardial SPECT in women and men. J Nucl Med. 1998 May;39(5):751-5. PMID 9591568
- [Background] Hachamovitch R, Berman DS, Kiat H, Bairey CN, Cohen I, Cabico A, Friedman J, Germano G, Van Train KF, Diamond GA. Effective risk stratification using exercise myocardial perfusion SPECT in women: gender-related differences in prognostic nuclear testing. J Am Coll Cardiol. 1996 Jul;28(1):34-44. doi: 10.1016/0735-1097(96)00095-2. PMID 8752792
- [Background] Pancholy SB, Fattah AA, Kamal AM, Ghods M, Heo J, Iskandrian AS. Independent and incremental prognostic value of exercise thallium single-photon emission computed tomographic imaging in women. J Nucl Cardiol. 1995 Mar-Apr;2(2 Pt 1):110-6. doi: 10.1016/s1071-3581(95)80021-2. PMID 9420775
- [Background] Hachamovitch R, Berman DS, Kiat H, Cohen I, Friedman JD, Shaw LJ. Value of stress myocardial perfusion single photon emission computed tomography in patients with normal resting electrocardiograms: an evaluation of incremental prognostic value and cost-effectiveness. Circulation. 2002 Feb 19;105(7):823-9. doi: 10.1161/hc0702.103973. PMID 11854122
- [Background] Galassi AR, Azzarelli S, Tomaselli A, Giosofatto R, Ragusa A, Musumeci S, Tamburino C, Giuffrida G. Incremental prognostic value of technetium-99m-tetrofosmin exercise myocardial perfusion imaging for predicting outcomes in patients with suspected or known coronary artery disease. Am J Cardiol. 2001 Jul 15;88(2):101-6. doi: 10.1016/s0002-9149(01)01601-0. PMID 11448403
- [Background] Shaw LJ, Hendel R, Borges-Neto S, Lauer MS, Alazraki N, Burnette J, Krawczynska E, Cerqueira M, Maddahi J; Myoview Multicenter Registry. Prognostic value of normal exercise and adenosine (99m)Tc-tetrofosmin SPECT imaging: results from the multicenter registry of 4,728 patients. J Nucl Med. 2003 Feb;44(2):134-9. PMID 12571200
- [Background] Marwick TH, Shaw LJ, Lauer MS, Kesler K, Hachamovitch R, Heller GV, Travin MI, Borges-Neto S, Berman DS, Miller DD. The noninvasive prediction of cardiac mortality in men and women with known or suspected coronary artery disease. Economics of Noninvasive Diagnosis (END) Study Group. Am J Med. 1999 Feb;106(2):172-8. doi: 10.1016/s0002-9343(98)00388-x. PMID 10230746
- [Background] Shaw LJ, Heller GV, Travin MI, Lauer M, Marwick T, Hachamovitch R, Berman DS, Miller DD. Cost analysis of diagnostic testing for coronary artery disease in women with stable chest pain. Economics of Noninvasive Diagnosis (END) Study Group. J Nucl Cardiol. 1999 Nov-Dec;6(6):559-69. doi: 10.1016/s1071-3581(99)90091-0. PMID 10608582
- [Background] Shaw LJ, Olson MB, Kelsey SF, et al. Using estimated functional capacity to optimize stress testing for diagnosis and prognosis of coronary artery disease in symptomatic women: Results from the NHLBI-sponsored Women Ischemia Syndrome Evaluation study., in preparation
- [Background] Amanullah AM, Kiat H, Friedman JD, Berman DS. Adenosine technetium-99m sestamibi myocardial perfusion SPECT in women: diagnostic efficacy in detection of coronary artery disease. J Am Coll Cardiol. 1996 Mar 15;27(4):803-9. doi: 10.1016/0735-1097(95)00550-1. PMID 8613606
- [Background] Amanullah AM, Berman DS, Hachamovitch R, Kiat H, Kang X, Friedman JD. Identification of severe or extensive coronary artery disease in women by adenosine technetium-99m sestamibi SPECT. Am J Cardiol. 1997 Jul 15;80(2):132-7. doi: 10.1016/s0002-9149(97)00306-8. PMID 9230147
- [Background] Hendel RC, Chen MH, L'Italien GJ, Newell JB, Paul SD, Eagle KA, Leppo JA. Sex differences in perioperative and long-term cardiac event-free survival in vascular surgery patients. An analysis of clinical and scintigraphic variables. Circulation. 1995 Feb 15;91(4):1044-51. doi: 10.1161/01.cir.91.4.1044. PMID 7850940
- [Background] Heller GV, Herman SD, Travin MI, Baron JI, Santos-Ocampo C, McClellan JR. Independent prognostic value of intravenous dipyridamole with technetium-99m sestamibi tomographic imaging in predicting cardiac events and cardiac-related hospital admissions. J Am Coll Cardiol. 1995 Nov 1;26(5):1202-8. doi: 10.1016/0735-1097(95)00329-0. PMID 7594033
- [Background] Amanullah AM, Berman DS, Erel J, Kiat H, Cohen I, Germano G, Friedman JD, Hachamovitch R. Incremental prognostic value of adenosine myocardial perfusion single-photon emission computed tomography in women with suspected coronary artery disease. Am J Cardiol. 1998 Sep 15;82(6):725-30. doi: 10.1016/s0002-9149(98)00463-9. PMID 9761081
- [Background] Elliott MD, Holly TA, Leonard SM, Hendel RC. Impact of an abbreviated adenosine protocol incorporating adjunctive treadmill exercise on adverse effects and image quality in patients undergoing stress myocardial perfusion imaging. J Nucl Cardiol. 2000 Nov-Dec;7(6):584-9. doi: 10.1067/mnc.2000.108737. PMID 11144473
- [Background] Samady H, Wackers FJ, Joska TM, Zaret BL, Jain D. Pharmacologic stress perfusion imaging with adenosine: role of simultaneous low-level treadmill exercise. J Nucl Cardiol. 2002 Mar-Apr;9(2):188-96. doi: 10.1067/mnc.2002.119973. PMID 11986564
- [Background] Thomas GS, Prill NV, Majmundar H, Fabrizi RR, Thomas JJ, Hayashida C, Kothapalli S, Payne JL, Payne MM, Miyamoto MI. Treadmill exercise during adenosine infusion is safe, results in fewer adverse reactions, and improves myocardial perfusion image quality. J Nucl Cardiol. 2000 Sep-Oct;7(5):439-46. doi: 10.1067/mnc.2000.108030. PMID 11083192
- [Background] Holly TA, Satran A, Bromet DS, Mieres JH, Frey MJ, Elliott MD, Heller GV, Hendel RC. The impact of adjunctive adenosine infusion during exercise myocardial perfusion imaging: Results of the Both Exercise and Adenosine Stress Test (BEAST) trial. J Nucl Cardiol. 2003 May-Jun;10(3):291-6. doi: 10.1016/s1071-3581(02)43236-9. PMID 12794628
- [Background] Gibbons RJ, Chatterjee K, Daley J, Douglas JS, Fihn SD, Gardin JM, Grunwald MA, Levy D, Lytle BW, O'Rourke RA, Schafer WP, Williams SV. ACC/AHA/ACP-ASIM guidelines for the management of patients with chronic stable angina: executive summary and recommendations. A Report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Committee on Management of Patients with Chronic Stable Angina). Circulation. 1999 Jun 1;99(21):2829-48. doi: 10.1161/01.cir.99.21.2829. No abstract available. PMID 10351980
- [Background] Diamond GA, Forrester JS. Analysis of probability as an aid in the clinical diagnosis of coronary-artery disease. N Engl J Med. 1979 Jun 14;300(24):1350-8. doi: 10.1056/NEJM197906143002402. PMID 440357
- [Background] Chaitman BR, Bourassa MG, Davis K, Rogers WJ, Tyras DH, Berger R, Kennedy JW, Fisher L, Judkins MP, Mock MB, Killip T. Angiographic prevalence of high-risk coronary artery disease in patient subsets (CASS). Circulation. 1981 Aug;64(2):360-7. doi: 10.1161/01.cir.64.2.360. PMID 7249303
- [Background] Gibbons RJ, Balady GJ, Bricker JT, Chaitman BR, Fletcher GF, Froelicher VF, Mark DB, McCallister BD, Mooss AN, O'Reilly MG, Winters WL, Gibbons RJ, Antman EM, Alpert JS, Faxon DP, Fuster V, Gregoratos G, Hiratzka LF, Jacobs AK, Russell RO, Smith SC; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. Committee to Update the 1997 Exercise Testing Guidelines. ACC/AHA 2002 guideline update for exercise testing: summary article. A report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Committee to Update the 1997 Exercise Testing Guidelines). J Am Coll Cardiol. 2002 Oct 16;40(8):1531-40. doi: 10.1016/s0735-1097(02)02164-2. No abstract available. PMID 12392846
- [Background] Cerqueira MD, Weissman NJ, Dilsizian V, Jacobs AK, Kaul S, Laskey WK, Pennell DJ, Rumberger JA, Ryan T, Verani MS; American Heart Association Writing Group on Myocardial Segmentation and Registration for Cardiac Imaging. Standardized myocardial segmentation and nomenclature for tomographic imaging of the heart. A statement for healthcare professionals from the Cardiac Imaging Committee of the Council on Clinical Cardiology of the American Heart Association. Circulation. 2002 Jan 29;105(4):539-42. doi: 10.1161/hc0402.102975. No abstract available. PMID 11815441
- See also: Click here for more information about Midwest Heart Foundation — http://www.midwestheart.org